CLINICAL TRIAL: NCT05508945
Title: Silk Scaffold Surgical Incision Dressing Interventional Study
Brief Title: Silk Scaffold Surgical Incision Dressing
Acronym: SSSID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mehrdad Mark Mofid (Other)
Responsible Party: Sponsor-Investigator, Mehrdad Mark Mofid, Principal Investigator, San Diego Skin, Inc.
Organization: San Diego Skin, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSSID; 20204292 (Other: WCG IRB)
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Surgical Incision
Keywords: surgical incision dressing; surgical wound dressing; wound coverage; wound dressing; silk; contact dermatitis; SERI scaffold
MeSH Terms: conditions — Surgical Wound; Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: subjects receive 50% surgical incision coverage with experimental silk/adhesive prototype and 50% surgical incision coverage with FDA approved Dermabond Prineo OR FDA approved Steri-Strip.
Masking Description: Participants are not informed which dressing is Dermabond Prineo and which is SERI scaffold with dermaFLEX adhesive. Participants are informed they will be receiving both interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surgical Incision (Experimental): Abdominoplasty Surgical Incision, Breast Reduction Surgical Incision, Mastopexy Surgical Incision, or Belt Lipectomy Surgical Incision
  Interventions: Device: Dermabond Prineo Skin Closure System; Device: silk; Device: 3M Steri-Strip

INTERVENTIONS:
Device: Dermabond Prineo Skin Closure System — synthetic mesh patch is positioned and lightly pressed over 50% of the surgical incision. 2-octyl cyanoacrylate liquid adhesive is evenly applied over the mesh and allowed to dry
Device: silk — SERI surgical scaffold with dermaFLEX backing is positioned over the remaining 50% of the surgical incision
  Other Names: SERI surgical scaffold
Device: 3M Steri-Strip — non-woven rayon with adhesive backing is applied to 50% of the surgical incision.

SUMMARY:
Interventional Study of the novel clinical application of SERI surgical silk scaffold affixed with dermaFLEX medical adhesive as a wound dressing, compared to two separate current standard of care for surgical incision closure devices: Prineo Dermabond and 3M Steri-Strip. Both components of the silk wound dressing prototype are FDA approved materials for other indications. This study seeks to gain insight of functionality of silk as a wound coverage material and determine variations of clinical outcomes in comparison to the synthetic mesh/cyanoacrylate device (Prineo Dermabond) and the nonwoven rayon/acrylate device (3M Steri-Strip) commonly implemented as a surgical wound dressing.

DETAILED DESCRIPTION:
Participants for the study will be selected from a population of patients who have voluntarily sought out and consented to cosmetic and/or reconstructive surgery performed by M. Mark Mofid M.D. Patients who request and consent to procedures named in the protocol will be considered for eligibility of participation. Dr. Mofid will make the final determination after a thorough clinical evaluation of the patients medical information. Participants undergoing procedures that result in a single continuous surgical incision will receive the either Prineo Dermabond closure device or 3M Steri-Strip surgical incision closure device on 50% of the surgical incision, and the SERI Scaffold/ dermaFLEX combination on the remaining 50% of the incision. An automated randomization app will be used to determine which side, left or right, will receive each dressing. For an abdominoplasty, the incision typically extends from hip to hip, across the lower abdomen. For this procedure, the Prineo Dermabond or 3M Steri-Strip will be applied from the center of the incision: the belly button, and to the end of the incision, or hip, of the randomly determined side. The SERI Scaffold and dermaFLEX adhesive will be placed on the opposite side of the incision. For procedures that result in separate incisions, such as Breast Reductions, one breast will receive the Prineo Dermabond or 3M Steri-Strip coverage, while the other breast will receive the SERI Scaffold w/ dermaFLEX coverage. The sides will be determined through an automated randomization app. The surgeon, Dr. Mofid, will be informed which side will receive each dressing immediately before the respective dressings are to be applied. The dressings will subsequently be compared and evaluated during post-operative visits. Participants will complete a questionnaire at each designated post-operative visit and answers will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit fluency and literacy in English
* Exhibit adequate cognitive ability to consent to experimental research
* Ability to obtain pre-operative clearance from an unaffiliated primary care physician prior to surgery as deemed necessary under M. Mark Mofid's predetermined standard of care guidelines for patients

Exclusion Criteria:

* Diagnosis of autoimmune disorders
* Diagnosis of allergy to DERMABOND Topical Skin Adhesive, STERI-STRIP skin closure strips, polyester mesh, and/or silk
* Any acute or chronic condition that may inhibit ability to participate in the full duration of study
* Inability to give informed consent
* Investigator decision that subject is no a suitable candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-08-19 (Actual)

PRIMARY OUTCOMES:
Presence of Contact Dermatitis | 3 days post operation, 7 days post operation, 14 days post operation, 28 days post operation, 42 days post operation
  Participants will self report symptoms of Contact Dermatitis surrounding the treated area quantified on a scaling system of 0-10 based upon the following criteria: Skin Discomfort, Skin Irritation, and Skin Itching.
  The Principal Investigator will determine the clinical appearance of Contact Dermatitis surrounding the treated area quantified on a scaling system of 0-10 based upon the following criteria: Skin Rash and Skin Redness

SECONDARY OUTCOMES:
Wound Dressing Detachment | 3 days post operation, 7 days post operation, 14 days post operation
  Participants will be evaluated by the Principal Investigator for signs of detached or displaced wound dressings. Participants will self report spontaneous detachment of wound dressing prior to anticipated dressing removal, scheduled 14 days post-operation. The results will be quantified by a measure of "Yes" or "No".

OTHER OUTCOMES:
Presence of Infection | 3 days post operation, 7 days post operation, 14 days post operation, 28 days post operation, 42 days post operation
  The Principal Investigator will evaluate presence of infection at the surgical site based upon the standard clinical evidence of infection. The results will be quantified by a measure of "Yes" or "No".

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Mark Mofid, M.D., Principal Investigator — San Diego Skin
Locations (1):
- San Diego Skin, Inc., La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Informed Consent Form will be shared upon completion of trial. Statistical Analysis Plan and Clinical Study Report will be made available 6 months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 1 year after publication.

REFERENCES:
- See also: Silkworm silk-based materials and devices generated using bio-nanotechnology — https://pubs.rsc.org/en/content/articlelanding/2018/CS/C8CS00187A